CLINICAL TRIAL: NCT06325020
Title: ORACLE: Objective Risk Assessment in Patients With Possible Anginal Chest Pain Using Leading Technology
Brief Title: Objective Risk Assessment in Patients With Possible Anginal Chest Pain Using Leading Technology
Acronym: ORACLE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 337367
Record Dates: First submitted 2024-03-06; First posted 2024-03-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Angina, Stable; Coronary Artery Disease
Keywords: angina, chest pain, cardiac troponin, risk stratification
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Angina Pectoris; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be taken from participants, with their consent, and stored to allow for future biomarker exploration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with possible angina: Participants will complete a digital health questionnaire, at home, that asks about their risk factors for coronary artery disease, past medical history and their symptoms.
  Patients will then have a standard 12 lead ECG and perform their own personal ECG. They will then have high sensitivity cardiac troponin measured.
  The results of all of the above will allow patients to be started as low, intermediate or high risk for future cardiovascular events.
  Interventions: Other: The assessment of patients with possible angina using the ORACLE pathway

INTERVENTIONS:
Other: The assessment of patients with possible angina using the ORACLE pathway — Participants will complete a digital health questionnaire, at home, that asks about their risk factors for coronary artery disease, past medical history and their symptoms.
  Patients will then have a standard 12 lead ECG and perform their own personal ECG. They will then have high sensitivity cardiac troponin measured.
  The results of all of the above will allow patients to be started as low, intermediate or high risk for future cardiovascular events.

SUMMARY:
The ORACLE study is an observational cohort study designed to explore the feasibility of providing an assessment of chest pain for patients with suspected angina within one working day of referral to specialist services.

The primary objective is to determine the feasibility of delivering an objective assessment of risk for participants who have been referred by their primary care provider to the rapid access chest pain clinic with possible angina in a community setting using point of care and patient facing technologies within one working day of referral.

Participants will complete a digital health questionnaire, at home, that asks about their risk factors for coronary artery disease, past medical history and their symptoms.

Patients will then have a standard 12 lead ECG and perform their own personal ECG. They will then have high sensitivity cardiac troponin measured by point of care high sensitivity cardiac troponin assays as well as a core lab assay.

The results of all of the above will allow patients to be started as low, intermediate or high risk for future cardiovascular events.

DETAILED DESCRIPTION:
Recent onset of angina is a clinical manifestation of unstable or progressive coronary artery disease and is a common presentation within primary care. Evaluation can be challenging as access to objective measures of risk and diagnostic testing are limited in this setting. Due to capacity, not all patients referred to the rapid access chest pain clinic can be reviewed within this clinic.

Patients are often high risk with suspected obstructive coronary artery disease, and the aim should be for review, assessment and if required, initiation of therapy, without undue delay.

This study has been designed to explore the feasibility of delivering a virtual chest pain assessment for patients with new onset chest pain. It is an observational cohort study, that uses a combination of digital tools to capture relevant patient information and clinical history, point-of-care high-sensitivity cardiac troponin testing and electrocardiography.

This pathway will aim to provide an objective assessment of risk on the next working day following primary care contact to all patients referred to the rapid access chest pain clinic.

On completion of this assessment patients will be stratified to low, intermediate or high risk groups based on their symptoms, risk factors, point of care troponin value (ng/l) and ECG. The results will not be made available to the clinical team unless the patients was at risk of harm (acute coronary syndrome or arrhythmia). Patients will return to receive routine clinical care.

The investigators plan to recruit 300 participants or for six months, whatever arises first. Participants can only be recruited once during the study period.

ELIGIBILITY:
Inclusion Criteria:

* >30 years of age
* Referral to the rapid access chest pain clinic with possible new onset or worsening angina

Exclusion Criteria:

* Inability to give informed consent.
* Previous recruitment to the study.
* Acute coronary syndrome within 3 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the rapid access chest pain service within NHS Lothian will be eligible to participate in our feasibility study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in whom a chest pain risk assessment is complete within one working day of referral. | This is the time from referral to rapid access chest pain clinic through to completion of their visit, anticipated to be between 1 and 3 days.
  The proportion of participants who have been referred by their primary care provider to the rapid access chest pain clinic with possible angina in whom a complete risk assessment is delivered in a community setting using point of care and patient facing technologies within one working day of referral.

SECONDARY OUTCOMES:
Proportion of patients who can have their risk assessment completed in one, two or three or more working days from referral to service until completion of risk assessment. | This is the time from referral to rapid access chest pain clinic through to completion of their visit, anticipated to be between 1 and 3 days.
  The proportion of participants who have been referred by their primary care provider to the rapid access chest pain clinic with possible angina in whom a complete risk assessment is delivered in a community setting using point of care and patient facing technologies within one, two or three or more working days of referral.
Proportion of valid and interpretable point-of-care troponin tests | This will be completed during the patients study visit, anticipated to last 1 hour
  This will be the proportion of patients in whom a valid high sensitivity cardiac troponin result can be obtained from undertaking the point of care assay.
Proportion of personal electrocardiograms that are interpretable | This will be completed during the patients study visit, anticipated to last 1 hour
  This will be the proportion of patients in whom an interpretable personal ECG has been performed
Proportion of participants stratified as low, intermediate, or high risk using objective risk stratification. | This will be completed during the patients study visit, anticipated to last 1 hour
  This will be the proportion of patients who are stratified into low, intermediate or high risk groups on completion of their risk assessment.
Proportion of participants with and without a clinical diagnosis of angina stratified as low, intermediate, or high risk and according to triage status. | This will be obtained at 3 months following completion of the patient's assessment.
  This will be the proportion of patients who do and do not receive a clinical diagnosis of angina and this will be stratified by triage status
Proportion of participants with unscheduled Emergency Department attendance(s) at 3 months stratified as low, intermediate, or high risk and according to triage status. | This will be obtained at 3 months following completion of the patient's assessment.
  This will be the proportion of patients who present acutely to the emergency department in the 3 months following assessment. This will be stratified by risk stratification and their clinical triage status.
Proportion of participants with cardiac death or non-fatal myocardial infarction at 3 months stratified as low, intermediate, or high risk and according to triage. | This will be obtained at 3 months following completion of the patient's assessment.
  This will be the proportion of patients who have cardiac death or fatal myocardial infarction in the 3 months following assessment. This will be stratified by risk stratification and their clinical triage status.

OTHER OUTCOMES:
Proportion of participants reclassified as low, intermediate, or high risk using standard laboratory assays compared to point-of-care high-sensitivity cardiac troponin assay. | This will be completed during the patients study visit, anticipated to last 1 hour
  Patients will have a point of care troponin and a core laboratory high sensitivity troponin. The proportion of patients who are re-classified by the current laboratory clinical standard will be recorded
Proportion of participants reclassified as low, intermediate, or high risk using standard 12-lead compared to personal 12-lead electrocardiography | This will be completed during the patients study visit, anticipated to last 1 hour
  Patients will have a standard 12 lead and personal ECG. The proportion of patients who are re-classified by the current clinical standard 12 lead ECG will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDermott, MBCHB, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No